CLINICAL TRIAL: NCT00690417
Title: Vitamin D Inadequacy: Documentation in Rural Populations and Evaluation of Correction by Food Supplementation (Phase III; Manitowoc Prevalence Study)
Brief Title: Vitamin D Inadequacy in Rural Populations, Evaluation of Correction by Food Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-0211
Record Dates: First submitted 2008-01-07; First posted 2008-06-04 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Vitamin D Insufficiency; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)
- 2. 2500 IU vitamin D in a food preparation (Active Comparator): Daily ingestion of 2500 IU vitamin D in a food preparation.
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (vitamin D3) — low calorie (~60 calories) cookie-like disc containing 2,500 IU of vitamin D3, taken by mouth daily for 4 months

SUMMARY:
The purpose of the research is to describe vitamin D levels and bone status in a rural Wisconsin population. It is probable that individuals of varying age and ethnicity require different amounts of D to achieve optimal status. These likely scenarios will be explored in various populations. We hypothesize that the increase in serum 25(OH)D resulting from daily D3 ingestion is less pronounced with advancing age and different in Native than Caucasian Americans. In addition, the women in the middle age group, between the ages of 55 and 65, will have ultrasound tests completed to assess the impact of the Vitamin D supplementation on cardiovascular health.

ELIGIBILITY:
Inclusion criteria:

* Healthy, community-dwelling ambulatory women.
* Able and willing to sign informed consent.
* Ages: 20-30, 55-65 or >75
* Baseline serum 25OHD concentration > 10 ng/ml and < 60 ng/ml
* Not pregnant
* Willing to avoid use of cod-liver oil and non-study vitamin D supplementation; standard multiple vitamins containing ≤ 400 IU used no more than once daily will be allowed.
* Willing to utilize sunscreen of SPF-15 or higher when sun exposure for more than 15 minutes is expected.

Exclusion criteria:

* Current hypercalcemia (serum calcium > 10.5 mg/dl) or untreated primary hyperparathyroidism.
* History of nephrolithiasis
* Baseline 24-hour urine calcium > 250 mg
* Known risk factors for hypercalcemia, e.g., malignancy, tuberculosis, sarcoidosis, Paget's disease.
* History of any form of cancer within the past five years with the exception of adequately treated squamous cell or basal cell skin carcinoma.
* Renal failure; defined as a calculated creatinine clearance (using the Cockroft-Gault approach) of ≤ 25 ml/minute.
* Severe end-organ disease, e.g., cardiovascular, hepatic, hematologic, pulmonary, etc., which might limit the ability to complete this study.
* Treatment with any drug known to interfere with vitamin D metabolism, e.g., phenytoin, phenobarbital.
* Known malabsorption syndromes, e.g., celiac disease, active inflammatory bowel disease, etc.
* Known allergy to chocolate.
* Use of medications known to alter bone turnover including bisphosphonates, estrogen, selective estrogen receptor modulators, parathyroid hormone, testosterone or calcitonin.
* Treatment with high dose vitamin D (≥ 50,000 IU weekly) or any active metabolites of vitamin D, e.g., calcitriol, within six months of screening.
* Use of tanning beds or salons or unwillingness to utilize sunscreen during periods of sun exposure of 15 minutes or longer.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
the primary outcome is the proportion of postmenopausal women with D inadequacy defined by current consensus as a serum 25(OH)D < 30 ng/ml. | 2.5 years

SECONDARY OUTCOMES:
Prevalence of Vitamin D insufficiency in rural populations and ethnic differences in response to vitamin D supplementation | 2.5 year
The relationship between vitamin D supplementation and cardiovascular disease. | 2.5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Principal Investigator — University of Wisconsin - Institute on Aging
Locations (1):
- University of Wisconsin Osteoporosis Clinical and Research Program, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Gepner AD, Ramamurthy R, Krueger DC, Korcarz CE, Binkley N, Stein JH. A prospective randomized controlled trial of the effects of vitamin D supplementation on cardiovascular disease risk. PLoS One. 2012;7(5):e36617. doi: 10.1371/journal.pone.0036617. Epub 2012 May 7. PMID 22586483